CLINICAL TRIAL: NCT04266015
Title: A Randomized Trial of Intraoperative Feeding to Ameliorate Catabolic Response in Free Flap Reconstruction Surgery for Head-and-neck Cancer Defect
Brief Title: Anabolic Effects of Intraoperative Feeding in Reconstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, Superintendent, professor, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRP71108N
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Fasting; Feeding, Time Restricted; Stress-related Problem; Head and Neck Neoplasms; Catabolic State; Hyperglycemia Stress; Muscle Wasting; Complication,Postoperative
MeSH Terms: conditions — Fasting; Intermittent Fasting; Head and Neck Neoplasms; Muscular Atrophy; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized double-blind controlled trial
Who Masked: Participant, Care Provider
Masking Description: Participants: patients will receive general anesthesia before intervention Care providers: surgeons will be masked of the treatment group during operation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients assigned to control group will not receive feeding via the nasogastric tube during operation
- Intraoperative feeding group (Experimental): Patients assigned to intraoperative feeding group will receive enteral nutrition formula via the nasogastric tube during operation
  Interventions: Dietary Supplement: Enteral nutrition formula

INTERVENTIONS:
Dietary Supplement: Enteral nutrition formula — Intervention group will receive nasogastric feeding with commercially available liquid enteral diet (250 ml/can, Kcal/ml, 10.4 g protein/can) during free flap reconstruction at feeding rates 10-30 ml/h.
  Arms: Intraoperative feeding group

SUMMARY:
Perioperative fasting remains a common clinical practice in surgical patients to prevent the development of postoperative anesthesia- and surgical-related complications. Clinical observational studies indicated that the combination catabolic effects resulted from prolonged perioperative fasting and profound surgical stress are likely to induce extensive protein catabolism, muscle breakdown and impaired glycemic control during postoperative phase, leading to the development of severe complications. Furthermore, prolonged gastrointestinal fasting is associated with microbial translocation that deteriorates the early recovery after surgery. This clinical trial anticipates in determining the beneficial effect of intraoperative feeding to improve intraoperative hemodynamics and enhance postoperative recovery due to attenuation of systemic catabolism and improvement of insulin sensitivity to glycemic control.

DETAILED DESCRIPTION:
Perioperative fasting remains a common clinical practice in surgical patients, aiming to prevent pulmonary aspiration during anesthesia induction, improve bowel preparation, and ameliorate the development of postoperative nausea/vomiting or other surgical-related complications. Major head-and-neck tumor excision and reconstruction surgery is one of the most time-consuming surgeries that usually takes more than 12 h to complete. In addition to the preoperative fasting and postoperative recovery time periods, most of these patients will be fasted for more than 24-36 h before they are fed via nasogastric tubes in the postoperative care units. The combination catabolic effects resulted from prolonged perioperative fasting and profound surgical stress are likely to induce extensive protein catabolism, muscle breakdown and impaired glycemic control during postoperative phase. These catabolic responses may lead to the development of post-operative surgical site infection, delayed wound healing, re-intervention, cardiac arrest, and death in diabetic and non-diabetic patients. Furthermore, prolonged gastrointestinal fasting is associated with dehydration, perturbed gut integrity/permeability (leaky gut) and microbial (bacterial) translocation that deteriorates the early recovery after reconstruction surgery. The aim of this clinical trial is to test the effect of intraoperative feeding in patients receiving head-and-neck tumor excision and reconstruction surgery, and anticipate that reduction of perioperative fasting time may improve intraoperative hemodynamics and enhance postoperative recovery due to attenuation of systemic catabolism and improvement of insulin sensitivity to glycemic control.

This single-center clinical trial will be undertaken in a randomized, double-blind, placebo-controlled fashion, in which patients with advanced head-and-neck tumor who are scheduled for extended tumor resection and free-flap reconstruction will be randomly assigned to receive control (no intraoperative feeding) or intraoperative feeding group. Feeding via the nasogastric (NG) tube will start after the establishment of tracheostomy and completion of tumor resection at fusion rate of 10-30 ml/h (feeding diet 1 Kcal/ml and 0.04 g protein/ml). This trial anticipates in detecting differences in intraoperative hemodynamic stability and development of major postoperative complications, including delayed wound healing, surgical site infections and insulin-resistant hyperglycemia between controls and intraoperative feeding group. The outcomes of this clinical trial may provide fundamental evidence for vigorous enteric nutrition and energy support during prolonged high surgical stress operation.

ELIGIBILITY:
Inclusion Criteria:

* Advanced head-and-neck cancer
* Requires radical resection, tracheostomy and free flap reconstruction surgery

Exclusion Criteria:

* Anticipated total operation time < 6h
* Emergency operation
* Bowel obstruction
* Starts nasogastric feeding before operation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Number of participants that have reconstruction flap failure after operation | 7 days after free flap reconstruction
  The definition of flap failure includes vascular occlusion of flap, surgical wound infection or poor healing that requires surgical reintervention

SECONDARY OUTCOMES:
Number of participants that have perioperative complications | Start of free flap reconstruction surgery to 28 days after operation
  The definition of composite perioperative complications during and after operation, include intraoperative hemodynamic stability (hypotension and requirement of inotropes), postoperative insulin sensitivity, glycemic control, skeletal muscle wasting, inflammatory cytokine profiles, length of hospital stay, re-intervention, other postoperative complications, mortality during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Fuh Lam, MD, PhD, Principal Investigator — E-Da Hospital, Taiwan
Locations (1):
- E-Da Hospital, Yanchao, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Hwang TZ, Wang YM, Jeng SF, Lee YC, Chen TS, Su SY, Huang CC, Lam CF. Intraoperative Enteral Nutrition Feeding in Free-Flap Healing after Reconstruction Surgery for Head and Neck Cancers. Otolaryngol Head Neck Surg. 2023 Oct;169(4):843-851. doi: 10.1002/ohn.335. Epub 2023 Mar 24. PMID 36960779